CLINICAL TRIAL: NCT05365412
Title: Clinicopathological Characteristics of Colon Cancer in Young Age
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1901-514-112
Record Dates: First submitted 2022-04-24; First posted 2022-05-09 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Colo-rectal Cancer; Molecular Pathway Deregulation
Keywords: colorectal cancer; prognosis; sex difference
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Microinstability (MSS, MSI-L, MSI-H), DNA mismatch repair genes (hMLH1, hMSH2, hMSH6, hPMS2), RAS genes (KRAS, NRAS, HRAS), BRAF mutations from cancer tissue will be analyzed using immunohistochemistry (IHC) and reverse transcriptase polymerase chain reaction (RT-PCR).
  In addition, the expression of estrogen and androgen receptors will further be analyzed in each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Colorectal cancer group: Patients treated after being diagnosed with colorectal cancer

SUMMARY:
A Study on the Characteristics of Colorectal Cancer by Age and sex.

DETAILED DESCRIPTION:
The investigators aimed to investigate the prognosis according to sex and age by analyzing the clinical, pathophysiological, and molecular characteristics of colorectal cancer (CRC), and to find the factors influencing the prognosis of CRC.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated after being diagnosed with colorectal cancer

Exclusion Criteria:

* Patients under age of 18 years, or patients who cannot choose whether to participate or not
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated after being diagnosed with colorectal cancer, and agreed to participate
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Survival (overall/disease-specific) according to sex, molecular profiles and sex hormone receptors | From date of enrollment until the date of death from colorectal cancer or from any cause, assessed up to 120 months
  Time from diagnosis to death

SECONDARY OUTCOMES:
Disease-free survival according to sex, molecular profiles and sex hormone receptors | From date of enrollment until the date of first documented recurrence of colorectal cancer, assessed up to 120 months
  Time from diagnosis to recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, MD, PhD, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No